CLINICAL TRIAL: NCT02149810
Title: Automatic Self-transcending Meditation (ASTM) Therapy Versus Treatment as Usual (TAU) in Late Life Depression: Implications for Cardiovascular Health and Cross-fertilization Across Different Levels of Care.
Brief Title: Automatic Self Transcending Meditation Versus Treatment as Usual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Automatic Self Transcending Meditation and Treatment as Usual (Experimental): Participants in the ASTM group will undergo ASTM training in groups of four .This involves participating in four, 90-120 minutes sessions each of four consecutive days. This will be followed by once weekly 45-60 minute follow up sessions for 12 weeks. In addition participants will be asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants will be asked to log practice frequency and any other noteworthy observations in the log sheet provided to them.
  Interventions: Behavioral: Automatic Self Transcending Meditation
- Treatment as Usual (No Intervention): Participants randomized to control arm (TAU) will continue to receive their treatment as usual including antidepressant medications and/or psychotherapy

INTERVENTIONS:
Behavioral: Automatic Self Transcending Meditation — as above
  Other Names: ASTM
  Arms: Automatic Self Transcending Meditation and Treatment as Usual

SUMMARY:
Depression is a leading contributor to global burden of disease. Antidepressants do not provide adequate response for many patients. Mind-body therapies are often safe, increasingly embraced by patients, however good quality clinical trial data is limited. The PI has shown that there is autonomic instability in patients with late life depression (LLD). Through his team of across discipline researchers he will investigate benefits of one adjunctive mind-body intervention, automatic self transcending meditation on autonomic instability in LLD and depressive symptoms compared to treatment as usual. If results are positive, such an intervention could be used for management of LLD across all levels of care.

WHAT IS THE INNOVATION AND MAIN QUESTION/HYPOTHESIS UNDERLYING THIS PROPOSAL? The main study objectives are to assess heart rate variability (HRV), other autonomic parameters and depression scores in patients with late life depression undergoing an innovative mind-body therapy 'automatic self-transcending meditation' (ASTM) not previously evaluated in a randomized controlled manner in the treatment of late life depression.

It is expected that adding ASTM to TAU will be better than TAU in improving HRV, depression severity and other autonomic parameters in the treatment of LLD. It is expected that this intervention will produce significant anxiolytic and enhanced quality of life outcomes and will have no major side effects. If the results of this study are positive, it is possible that this intervention could be considered as treatment option for the management of this disabling illness in primary, secondary and tertiary care. Such treatment option would be more cost and staff effective, and self empowering than the current standard of care. It could also provide treatment options for patients who are currently resistant to their antidepressants.

DETAILED DESCRIPTION:
Late life depression and cardiovascular autonomic function:

Major depressive disorder in the elderly (in those >60 years of age), also known as late life depression (LLD), is common, disabling and associated with a high mortality rate caused by suicide as well as cardiovascular events compelling appropriate treatment. Research shows that in a naturalistic setting response rate to at least one antidepressant trial of adequate dose and duration alone is around 30-40% thereby necessitating usage of additional interventions. Such therapies include psychological therapies, and, recently, various forms of treatments loosely defined as mind-body therapies such as biofeedback, energy healing, meditation, guided imagery, and yoga. Mind-body therapies are being increasingly embraced by patients as they have negligible side effects, are easy to administer and display beneficial effects on the quality of life as well as comorbid anxiety. There is increasing research on the mechanisms and benefits of such therapies, however, good quality trial data is scant. It is well established that antidepressants work by mostly modifying neurotransmitter levels in the brain. On the other hand, some mind-body therapies target multiple organ systems and hence could offer neurobiological advantages as depression is now recognised as a multi-system disorder. This is particularly relevant to the LLD population where there is increased prevalence of comorbid cardiovascular disorders. Hence, some mind body therapies when offered in combination with antidepressants might have a beneficial effect on both depression and the cardiovascular system.

One of the ways of assessing the cardiovascular system is through measurement of various autonomic parameters i.e. heart rate, blood pressure and heart rate variability. The most commonly reported is heart rate variability (HRV) which is a manifestation of the interplay of the central nervous system and the autonomic nervous system on a beat-by-beat basis. One of the ways of its estimation is by calculating the elapsed time between two consecutive waves, called R waves, on a person's electrocardiogram (ECG). A consistent finding has been that there is reduced HRV in people who have suffered a myocardial infarction (MI), and this phenomena is a predictor of subsequent cardiac arrhythmia and even death. In addition, through previous work the PI has found that in LLD there are significant cardiovascular autonomic disturbances compared to age matched controls after controlling for various risk factors. Other studies conducted in depression across the human life span have found similar results. Hence, if there is a mind-body treatment that specifically targets autonomic dysfunction and has a positive benefit on depressive symptoms, it would be valuable to asses. The investigators would like to investigate such a therapy which has been selected based on previous reports of beneficial effects but has not been evaluated in a randomised controlled trial of LLD patients.

Automatic self-transcending meditation (ASTM):

ASTM is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness. Research suggests that ASTM is easier to learn and to teach in comparison to other meditation techniques including mindfulness. Studies of adult and elderly ASTM practitioners have documented reductions in depressive symptoms, as well as improvements in cardiovascular function among elderly with and without cardiovascular disease. A study of adults with CVD further demonstrated improvements in HRV. Research further suggests ASTM may be particularly well suited to elderly populations. In a randomized controlled trial of elderly retirement home residents which evaluated ASTM with two other meditative techniques and treatment as usual, ASTM produced significantly greater improvements in cognitive function, cardiovascular function and quality of life than all other treatment conditions. A subsequent meta-analysis of all-cause mortality rates among hypertensive elderly who had participated in stress reduction interventions found that ASTM practitioners had a 30% lower cardiovascular mortality rate than four other meditative or relaxation interventions.

The investigators predict that ASTM augmentation is an effective intervention that ameliorates the autonomic disturbance associated with LLD, and possibly has beneficial effects on depressive symptoms as compared to a control treatment as usual (TAU) group.

Primary hypothesis: The investigators hypothesise that in patients with LLD, ASTM+TAU will lead to a significant increase in HRV from baseline to end of study period as compared to TAU.

Secondary hypotheses: The investigators hypothesise that ASTM+TAU will cause a) significant fall in depression scores b) significant improvement in other autonomic parameters including heart rate and blood pressure changes in presence of a physiological stress test (hand grip) c) significant improvement in depression related symptom pathologies including impaired quality of life and anxiety; compared to TAU.

Study Design:

This study is a single-centre, single blind longitudinal randomized controlled naturalistic trial. Research participants will be 96 men and women (48 in each group), 60-85 years of age, who have mild to moderate major depressive disorder (MDD). Participants will be recruited from primary, secondary and tertiary care centres in London, Ontario.

Study recruitment:

It is expected that the study will recruit from primary secondary and tertiary care practices in London identified by the investigators at a rate of at least 2 participants per week over a period of 76 weeks allowing attainment of a sample size of n=96. Advertisements about the study will be placed at key areas around the city including various community centres and libraries.

Usual standard of care at the trial site:

The standard of care for patients with late life depression involves starting them on an appropriate antidepressant from various classes such as SSRIs, (fluoxetine, fluoxamine, paroxetine, citalopram, escitalopram, sertraline, paroxetine), or NaSSA (mirtazapine) or Bupropion. Patients are also prescribed additional anxiolytic medications like benzodiazepines and trazodone if deemed necessary. Participants will be initiated and maintained on appropriate dosages of such medications as part of standard of care. The psychiatrist and/or his multidisciplinary team members might offer supportive therapy as part of standard of care.

Screening and initial assessments:

Potential participants will be screened as per inclusion and exclusion criteria. Upon selection, the following scales will be administered: interview for comorbid medical conditions (Cumulative illness rating scale- Geriatrics, CIRS-G), a screening cognitive examination (Mini Mental State Examination (MMSE)), depression severity assessment (Hamilton Rating Scale for Depression score (HRSD 17 items), Clinical Global Impression (CGI), self rated Geriatric Depression Scale (GDS)), anxiety (Geriatric Anxiety Inventory (GAI)), side effects (Toronto Side Effects Scale, (TSES)), Quality of Life (QOL profile seniors version (QOLPS), physical activity assessment (Physical activity scale of the elderly, PASE questionnaire).

Randomization:

Participants will be randomized to either ASTM+TAU or TAU equally (1:1) using computer generated randomisation numbers available at random.org. Concealment of randomisation will be ensured by independent staff performing randomisation.

Medication adherence follow-up:

All medication types will be permitted in this study. Any dosage modifications will be recorded.

Measurement of outcomes:

PRIMARY (HEART RATE VARIABILITY): Participants from both arms will be asked to report to the Laboratory for Brain and Heart Health at Western University Campus. Participants in both study arms will be requested to attend appointments at weeks 0 and 12 while participants in the ASTM arm will be requested to attend an additional assessment at 24 weeks.

1. Heart rate will be monitored using an electrocardiogram (ECG) with three adhesive leads.
2. Blood pressure will be measured using a small cuff placed on a finger (Finometer) or using a wrist cuff device (Colin Pilot). These continuous measures of blood pressure will be confirmed against values obtained periodically by an automated sphygmomanometer (Dinamap).
3. Electrocardiogram: A standard electrocardiogram will be collected via small surface electrodes on the chest to determine heart rate.
4. A bellows placed around the chest will provide information on respiratory excursions.

SECONDARY OUTCOME MEASURES:

Depression and comorbid symptoms will be assessed by a blinded rater on various scales at study visit days (week 0, 4, 8, and 12 for all participants and ASTM participants will attend an additional assessment at week 24). These scales are the rater assessed (Hamilton Rating Scale for Depression score (HRSD 17 items)) and Clinical Global Impression (CGI). Self rated scales include the Geriatric Depression Scale (GDS)), anxiety (Geriatric Anxiety Inventory (GAI)), Physical activity (PASE), adverse events (TSES) and quality of life (QOLPS).

Statistical analysis plan:

The main outcome of interest, HRV, will be calculated by standard deviation of all R-R intervals (SDNN) on ECG, root-mean square of successive differences (RMSSD), and number of R-R intervals differing by >50 m sec from adjacent intervals (NN50) in time domain analysis.

Analyses will be conducted on a PC running SAS v9.4 (SAS Institute Inc. Cary, USA) on a Windows 7 Platform. Demographic and clinical characteristics of the intervention (SSM) and control (TAU) condition will be compared by independent samples t-tests and χ2 or Fisher's exact test for continuous and categorical data, respectively. Linear mixed models (described below), controlling for baseline score, will be used to compare the SSM and TAU groups' change score from baseline to 12-week follow-up on SDNN and LF HRV (primary outcome) and depression severity (HRSD-17) (secondary outcome). Other exploratory outcomes will be evaluated in a similar way. Linear mixed models will also be used to compare the percent change in HRSD-17 scores, whereas generalised linear models will be used to compare the proportion of patients who responded to the intervention (≥50% decrease from baseline on the HRSD, defined a priori) and the proportion of patients who achieved remission (scores ≤7 on the HRSD-17, defined a priori) at the end of intervention (week 12). Linear mixed models with variance components covariance structure will be used in comparing HRSD-17 scores between groups (SSM and TAU), time (week 0, 4, 8 and 12) and group × time interaction. All HRV-related measures will be natural log-transformed. Cohen's d will be calculated by dividing the mean difference in change scores between the two groups by the s.d. of the control groups' change score. Following established guidelines, the linear mixed models will account for the partially nested design, which allows clustering in the intervention group (because of participants experiencing a group-based intervention, added as a random effect) and no clustering in the control group. Using this method, different hierarchical structures can be fit for the two groups. PROC MIXED will be used for continuous outcome variables, and PROC GLIMMIX will be used for binary outcome variables. Restricted maximum likelihood estimates will be used and the d.f. adjusted with the Satterthwaite method. Residual and influence diagnostics will be checked to confirm if the models fit the data well. The level of statistical significance will be set at α = 0.05. Complete-case analysis will be used.

Interim analysis may be completed in order to meet one or more of these conditions a) funder reporting requirements and/or b) research training requirements of students and/or c) data safety monitoring for stop or continue decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Of either gender, between the age range of 60-85 years.
2. Have an Axis 1 diagnosis of mild to moderate major depressive disorder or bipolar disorder with HAMD-21 score of 8 to 22.
3. Consuming single agent or combination antidepressant therapy at therapeutic doses for a minimum of four weeks.
4. Of good general physical health with no severe cardiovascular disease in the past 12 months, no past history of neurological disease or seizures or history of diabetic neuropathy.
5. Sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 45 minutes.
6. Willing and able to attend 4 initial ASTM training sessions and 75% of weekly follow up sessions.

Exclusion Criteria:

1. Participating in other similar studies.
2. Other significant mental health diagnosis (including Dementia, Substance dependence, Post traumatic stress disorder, panic disorder, Obsessive compulsive disorder, dissociative disorder, neurocognitive disorder and Personality disorder)
3. High risk of suicide as elicited by clinical interview.
4. Psychotic episodes within the past 12 months.
5. Recent (within the past 6 months) head trauma that required emergency care
6. Currently practicing any type of formal meditation, mindfulness or breathing techniques. 7. patients with severe cardiovascular disease in the past 12 months (myocardial infarction, stroke or TIA) as well as history of neurological disease (including Parkinson's Disease) or seizures

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: akshya vasudev, MD, MRCPsych, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Amtul Z, Arena A, Hirjee H, Khan ZU, Maldeniya PM, Newman RI, Burhan AM, Wetmore S, Vasudev A. A randomized controlled longitudinal naturalistic trial testing the effects of automatic self transcending meditation on heart rate variability in late life depression: study protocol. BMC Complement Altern Med. 2014 Aug 19;14:307. doi: 10.1186/1472-6882-14-307. PMID 25134497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment strategy consisted of advertisements placed in community centers and libraries in London (Ontario, Canada)and surrounding areas, with the headline 'A Meditation Study for Seniors looking for Relief from Feeling Low and Depressed'. We screened 270 potential participants from June 2014 to August 2016, through physician referrals and recruitment posters. Of these, 95 met the study criteria and were enrolled and randomized.
Groups:
- Automatic Self Transcending Meditation and Treatment as Usual: Participants in the ASTM group underwent ASTM training in groups of four or more. This involved participating in four, 90-120 minute sessions each on four consecutive days. This was followed by once weekly 45-60 minute follow up sessions for 12 weeks. In addition participants were asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants were asked to log practice frequency and any other noteworthy observations in the log sheet provided to them.
- Treatment as Usual: Participants randomized to the control arm (TAU) continued to receive their treatment as usual including antidepressant medications and/or psychotherapy
Period: Overall Study
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Started | 48 | 47
Baseline | 47 | 44
Week 4 | 43 | 42
Week 8 | 40 | 43
Week 12 | 40 | 43
Week 24 | 31 | 0 (Not applicable study was amended such that week 24 data was not collected for TAU participants.)
Completed | 40 | 43
Not Completed | 8 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was completed only for those participants who completed a week 12 (primary end point) assessment.
Groups:
- Automatic Self Transcending Meditation and Treatment as Usual: Participants in the ASTM group underwent ASTM training in groups of four or more. This involved participating in four, 90-120 minutes sessions each of four consecutive days. This was followed by once weekly 45-60 minute follow up sessions for 12 weeks. In addition participants were asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants were asked to log practice frequency and any other noteworthy observations in the log sheet provided to them.
- Total: Total of all reporting groups
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.45 (5.80) | 68.30 (6.50) | 68.88 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 33 | 57
  Male | 16 | 10 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27 | 34 | 61
  Non-caucasian | 13 | 9 | 22
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.97 (5.00) | 30.81 (7.00) | 29.89 (6.00)
Mini Mental State Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini Mental State Exam (MMSE) is a cognitive function test for use in elderly patients. This exam includes tests of orientation, attention, memory, language and visual-spatial skills. Scores range from 0 to 30 with higher scores indicating better cognitive functioning.
  units on a scale | 28.55 (1.70) | 29.00 (1.40) | 28.78 (1.55)
Cumulative Illness Rating Scale for Geriatrics (CIRS-G) [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) compiles and quantifies medical problems in elderly patients. The CIRS-G rates different body systems from 0 to 4 with 0 indicating no problem, 1 current mild or past significant problem, 3 severe/constant significant disability/"uncontrollable" chronic problems, 4 extremely severe/immediate treatment required/end organ failure/severe impairment in function. A total is calculated for all body systems with scores ranging from 0 to 56, with lower scores indicating better health.
  units on a scale | 9.46 (3.80) | 8.53 (3.70) | 9.00 (3.75)
Late onset of Major Depressive Episode [Count of Participants; unit: Participants] — Late onset of a major depressive episode was defined as the first depressive episode occurring at the age of 50 or older. A count of the number of participants who self-reported their first depressive episode as occurring at age 50 or older is reported. Population: There were 7 cases of missing data for onset of major depressive episode.
  Participants
    number analyzed (Participants) | 37 | 39 | 76
    (all) | 23.00 | 25 | 48
Two or More Major Depressive Episodes [Count of Participants; unit: Participants] — Population: There were 8 cases of missing data for frequency of major depressive episodes.
  Participants
    number analyzed (Participants) | 36 | 39 | 75
    (all) | 25 | 26 | 51
Smoker [Count of Participants; unit: Participants] — Population: There were 12 case of missing data for smoking status.
  Participants
    number analyzed (Participants) | 33 | 38 | 71
    (all) | 4 | 6 | 10
Taking antidepressant medications [Count of Participants; unit: Participants] | 30 | 26 | 56
Greater than 1 alcohol drink per week [Count of Participants; unit: Participants] — Population: There were 11 cases of missing data for drinking status.
  Participants
    number analyzed (Participants) | 34 | 38 | 72
    (all) | 12 | 14 | 26
Greater than 1 alcohol drink per week [Count of Participants; unit: Participants] — Population: There were 11 cases of missing data for drinking status.
  Participants
    number analyzed (Participants) | 34 | 38 | 72
    (all) | 12 | 14 | 26
Taking two or more antidepressant medications [Count of Participants; unit: Participants] | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability (SDNN) From Baseline to End of Study
Description: autonomic measure of heart rate variability was assessed at baseline as well as at end of intervention (week 12).
Time Frame: Baseline and week 12
Population: Four participants were missing data for autonomic measures.
Measure: Mean (95% Confidence Interval); unit: S.D. of the normalized N-N interval
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 37 | 42
S.D. of the normalized N-N interval | -0.006 [-0.15 to 0.14] | -0.116 [-0.26 to 0.03]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; The primary focus of this study was the interaction effect of treatment on heart rate variability at Weeks 0 and 12. On the assumption that this effect size is medium (Cohen's f = .25), calculations (using G*Power) 23 indicate that a sample size of 80 yield power estimates of .99 for both the interaction and the main effect of time. The study enrolled 95 participants to account for participant attrition; Test type: Superiority; p = 0.28, Mixed Models Analysis — The a priori threshold for statistical significance was p = 0.05; Linear mixed models, controlling for baseline score, were used to compare the SSM and TAU groups' change score from baseline to 12-week on SDNN; Mean Difference (Net) = 0.109, 95% CI 2-sided [-0.09 to 0.31]

2. Primary Outcome: Change in Heart Rate Variability (Low Frequency HRV) From Baseline to End of Study
Description: autonomic measure of heart rate variability was assessed at baseline as well as at end of intervention (week 12).
Time Frame: Baseline and week 12
Population: Four participants were missing data for autonomic measures.
Measure: Mean (95% Confidence Interval); unit: msec^2
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 37 | 42
msec^2 | 0.017 [-0.32 to 0.35] | -0.017 [-0.36 to 0.33]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.89, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Linear mixed models, controlling for baseline score, were used to compare the SSM and TAU groups' change score from baseline to 12-week on LF HRV; Mean Difference (Net) = 0.034, 95% CI 2-sided [-0.44 to 0.51]

3. Secondary Outcome: Hamilton Rating Scale for Depression 17 Item
Description: Change in Hamilton 17 (HDSR-17) item depression rating scale from baseline to week 12. Minimum value is 0, maximum value is 52; lower values indicate better outcomes.
Time Frame: Baseline and at week 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | -3.96 [-6.00 to -1.91] | -1.30 [-2.65 to 0.05]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.030, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = -2.66, 95% CI 2-sided [-5.05 to -0.26]

4. Secondary Outcome: Geriatric Anxiety Inventory
Description: Change in geriatric anxiety inventory (GAI). Scores range from 0 to 20 with lower scores indicating a better outcome.
Time Frame: Baseline and week 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | -3.71 [-5.15 to -2.26] | -1.34 [-2.77 to 0.10]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.021, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = -2.37, 95% CI 2-sided [-4.37 to -0.36]

5. Secondary Outcome: Physical Activity Scale for the Elderly
Description: Change in physical activity scale for the elderly (PASE). Scores range from 0 to 400 or more, with higher scores indicating a better outcome.
Time Frame: Baseline and week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | 3.32 [-12.02 to 18.67] | -7.68 [-18.09 to 2.73]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.22, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = 11.00, 95% CI 2-sided [-7.01 to 29.01]

6. Secondary Outcome: Quality of Life Profile: Seniors Version (Brief)
Description: Change in quality of life profile seniors version (QOLPS) scale. Scores range from 0 to 90 with higher scored indicating a better outcome.
Time Frame: Baseline and week 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | 10.23 [2.95 to 17.50] | 8.31 [0.63 to 16.00]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.72, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = 1.91, 95% CI 2-sided [-8.54 to 12.37]

7. Secondary Outcome: Clinical Global Impression - Global Improvement Scale
Description: Change in Clinical Global Impression - Global Improvement Scale (CGI-I). Scores range from 0 to 7 with lower values indicating a better outcome.
Time Frame: Week 0 and week 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | 2.85 [2.30 to 3.40] | 3.65 [3.26 to 4.04]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.018, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = -0.80, 95% CI 2-sided [-1.46 to -0.15]

8. Secondary Outcome: Toronto Side Effects Scale
Description: Change in the Toronto Side Effects Scale (TSES). Scores Range from 31 to 775 or higher with lower scored indicating a better outcome.
Time Frame: Week 0 and week 12.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
units on a scale | -14.75 [-30.46 to 0.96] | -14.62 [-30.25 to 1.02]
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Test type: Superiority; p = 0.99, Mixed Models Analysis — The a priori threshold for statistical significance was set at p = 0.05; Mean Difference (Net) = -0.14, 95% CI 2-sided [-21.94 to 21.66]

9. Post Hoc Outcome: Percentage of Participants Achieving a Response Criterion Set at ≥50% Decrease From Baseline, on the Hamilton Rating Scale for Depression 17 Item (HDRS 17)
Description: The percentage of participants achieving a significant response to the study intervention. Response was defined as a decrease in score of 50% or more on the Hamilton Rating Scale for Depression 17 item (HDRS 17) from week 0 to week 12.
Time Frame: Week 0 and week 12
Measure: Number; unit: % of participants achieving response
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
% of participants achieving response | 30.0 | 11.6
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Generalised linear models were used to compare the proportion of participants who responded to the intervention (≥50% decrease from baseline on the HRSD, defined a priori) at the end of intervention (week 12); Test type: Superiority; p = 0.049, Regression, Linear — The a priori threshold for statistical significance was set at p = 0.05; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.01 to 10.53]

10. Post Hoc Outcome: Percentage of Participants Achieving Remission on the Hamilton Rating Scale for Depression 17 Item (HDRS-17)
Description: The percentage of participants achieving remission, defined as a participant achieving a HDRS-17 score less than or equal to 7 at week 12 follow up.
Time Frame: Week 12
Measure: Number; unit: % of participants achieving remission
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 40 | 43
% of participants achieving remission | 40.0 | 16.3
Statistical Analysis 1: Comparison: Automatic Self Transcending Meditation and Treatment as Usual; Generalised linear models were used to compare the proportion of the proportion of participants who achieved remission (scores ≤7 on the HRSD, defined a priori) at the end of intervention (week 12); Test type: Superiority; p = 0.040, Regression, Linear — The a priori threshold for statistical significance was set at p = 0.05; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.06 to 10.64]

ADVERSE EVENTS:
Arm/Group | Automatic Self Transcending Meditation and Treatment as Usual | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43

LIMITATIONS AND CAVEATS:
This study lacked an active comparator to control for variables such as instructor attention, socializing in a group atmosphere and leaving one's residence for the study intervention. Our study may have been underpowered to assess the HRV changes as well as the potential long-term cardiovascular beneficial effects of this intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT02149810/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02149810/ICF_001.pdf